CLINICAL TRIAL: NCT05298280
Title: Vertical Effects in Class II Patients Treated With Distalization: Comparison Between Multibracket Conventional Therapy and Clear Aligners
Brief Title: Vertical Effects in Class II Patients Treated With Distalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Roberta Lione, Associate Researcher, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 257/21
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Malocclusion, Angle Class II
Keywords: Class II; Pendulum; Distalization; Clear Aligners
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: Subjects enrolled in the study were randomly assigned to the two groups: Pendulum Group (PG) Clear Aligner Group (CAG). All subjects were treated by the same clinician.
  A computer-generated random number list was used to allocate patients to treatments. Block randomization was used to assign the same number of patients to each treatment. The allocation sequence was concealed by the statistician, who used opaque and sealed envelopes, sequentially numbered for each patient.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The observer (BA) who performed all the measurements was blinded to the group assignment. The study was blinded in regard to the statistical analysis: blinding was obtained by eliminating from the elaboration file every reference to patient group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pendulum Group (PG) (Active Comparator): In the PG, all patients received a pendulum appliance as described by Angelieri et al. The Nance button was anchored to the first and second premolars with removable wires.
  Interventions: Device: Pendulum appliance
- Clear Aligner Group (CAG) (Active Comparator): The treatment of sequential upper arch distalization was performed by the same board-certified orthodontists as proposed by Align Technology and described by Ravera et al.
  Interventions: Device: clear aligners

INTERVENTIONS:
Device: Pendulum appliance — In the PG, all patients received a pendulum appliance as described by Angelieri et al. The Nance button was anchored to the first and second premolars with removable wires. The 0.032-inch TMA wires were activated 45 degrees to produce a force of 200-250g per side. On average, intraoral reactivation of the distalizing springs was performed twice during the procedure. When a super Class I molar relationship was obtained, pendulum was replaced by a Nance holding arch. The average treatment duration was 8 months followed by bracket conventional therapy.
  Arms: Pendulum Group (PG)
Device: clear aligners — The standardized orthodontic intervention was represented by the maxillary molar distalization protocol proposed by Align Technology: it was planned in order to obtain a sequential distalization on the upper arch, and the staging was set at 0.25 mm per aligner. During sequential distalization aligners are set up to distalize one tooth at a time. The attachments were engineered by Align Technology to achieve predictable tooth movements. Each couple of aligners was worn for 7 days.
  Arms: Clear Aligner Group (CAG)

SUMMARY:
Class II malocclusion presents a major and common challenge to orthodontists. Treatment of Class II malocclusion is one of the most investigated and controversial issues in contemporary orthodontics because of the extensive variability of treatment strategies addressing the morphological characteristics of this malocclusion. The therapeutic approaches include tooth extractions, orthopedic appliances and extraoral or intraoral distalizing appliances. Maxillary molar distalization is one of the most common strategies to correct Class II molar relationship and it is commonly indicated for patients with maxillary dentoalveolar protrusion or minor skeletal discrepancies. One of the most used devices is Pendulum appliance, introducted by Hilgers in 1992.

In the last decades, the orthodontic treatment with removable clear aligners has become an increasing common choice because of the growing number of adult patients who ask for aesthetic and comfortable alternatives to conventional fixed appliances.

In 1997, Align Technology (Santa Clara, Calif) adapted and incorporated modern technologies to introduce the clear aligner treatment (CAT). Only few investigations have focused on the predictability of orthodontic tooth movement with CAT. A systematic review by Rossini et al. pointed out that among the dental movements analyzed in 11 studies, the bodily distalization was the most predictable.

Clinicians can consider the use of aligners in treatment planning for adult patients requiring 2 to 3 mm of maxillary molar distalization.

However, a detailed analysis of the skeletal and dental changes that compared pendulum appliance and clear aligners in class II treatment is still lacking.

On the basis of these considerations, the aim of the present prospective study was to analyze the effects on vertical dentoskeletal changes following maxillary molar distalization with pendulum and full fixed appliances and clear aligners.

DETAILED DESCRIPTION:
Class II malocclusion presents a major and common challenge to orthodontists. Treatment of Class II malocclusion is one of the most investigated and controversial issues in contemporary orthodontics because of the extensive variability of treatment strategies addressing the morphological characteristics of this malocclusion. The therapeutic approaches include tooth extractions, orthopedic appliances and extraoral or intraoral distalizing appliances. Maxillary molar distalization is one of the most common strategies to correct Class II molar relationship and it is commonly indicated for patients with maxillary dentoalveolar protrusion or minor skeletal discrepancies. One of the most used devices is Pendulum appliance, introducted by Hilgers in 1992. It is a tooth-tissue-borne appliance that includes a Nance button on the palate for intraoral anchorage and titanium-molybdenum coils that deliver a mild and continuous force to the maxillary molars. Despite its efficacy for maxillary molar distalization, there are side-effects, including labial/mesial tipping and protrusion of the maxillary incisors and premolars, distal tipping of the maxillary molars, increase in lower anterior face height, clockwise mandibular rotation, and extrusion of the first premolars. Consequently, these side-effects have to be corrected during the following fixed appliance treatment phase.

In the last decades, the orthodontic treatment with removable clear aligners has become an increasing common choice because of the growing number of adult patients who ask for aesthetic and comfortable alternatives to conventional fixed appliances.

In 1997, Align Technology (Santa Clara, Calif) adapted and incorporated modern technologies to introduce the clear aligner treatment (CAT). Only few investigations have focused on the predictability of orthodontic tooth movement with CAT. A systematic review by Rossini et al. pointed out that among the dental movements analyzed in 11 studies, the bodily distalization was the most predictable.

Simon et al. reported a high accuracy (88%) of the bodily movement of upper molars with aligners when a mean distalization movement of 2.7 mm was prescribed. The authors reported the best accuracy when the movement was supported by the presence of an attachment on the tooth surface. Furthermore, they underlined the importance of staging in the treatment predictability.

Ravera et al. showed that clear aligners are effective in distalizing maxillary molars in non-growing subjects without significant vertical and mesiodistal tipping movements. The authors reported that the lower facial height did not change at the end of the treatment. Therefore, clinicians can consider the use of aligners in treatment planning for adult patients requiring 2 to 3 mm of maxillary molar distalization.

However, a detailed analysis of the skeletal and dental changes that compared pendulum appliance and clear aligners in class II treatment is still lacking.

On the basis of these considerations, the aim of the present prospective study was to analyze the effects on vertical dentoskeletal changes following maxillary molar distalization with pendulum and full fixed appliances and clear aligners.

All subjects were selected according to the following inclusion criteria: bilateral Class II or end to end Class II molar relationship, skeletal Class I or II malocclusion (ANB angle between 2° and 7°), normodivergence on the vertical plane (SN^GoGn angle less than 37°), crowding in the lower arch (≤6 mm), good quality of pre and post treatment radiographs. All patients were in good general health with healthy periodontium, generalized probing depths not exceeding 3 mm, and no radiographic evidence of periodontal bone loss. The exclusion criteria were: patients who required functional appliance therapy, those who had previous orthodontic treatment or extraction, hypodontia, craniofacial syndromes or cleft, previous prosthodontic treatments of the upper molars.

A computer-generated random number list was used to allocate patients to treatments. Block randomization was used to assign the same number of patients to each treatment. The allocation sequence was concealed by the statistician, who used opaque and sealed envelopes, sequentially numbered for each patient. The observer (BA) who performed all the measurements was blinded to the group assignment. The study was blinded in regard to the statistical analysis: blinding was obtained by eliminating from the elaboration file every reference to patient group assignment.

Subjects enrolled in the study were randomly assigned to the two groups: Pendulum Group (PG) Clear Aligner Group (CAG)

The Pendulum Group (PG) consisted of 20 patients (15F, 5M) with a mean age of 17.2 ± 4.3 years. The Clear Aligners Group (CAG) comprised 20 patients (13F, 7M) with a mean age of 17.2 ± 3.2 years. Distalization's protocol in PG involved the activation of TMA wires till the achievement of Class I molar relationship. A protocol of sequential distalization was applied in the CAG. For each subject lateral cephalograms have been analyzed before treatment (T1) and at the end of the therapy (T2).

To determine the reliability of the method, 15 randomly selected radiographs were traced and digitized by the same investigator on two separate occasions at least 1 month apart. A paired t-test was used to compare the two measurements (systematic error). The magnitude of the random error was calculated by using the method of moment's estimator (MME) (32).

The primary outcome was considered the changes in total vertical dimension (SN^GoGn) while secondary outcome was considered reduced Overjet. Exploratory statistics revealed that all cephalometric variables were normally distributed (Kolmogorov-Smirnov test) with equality of variances (Levene's test).

Descriptive statistics and statistical between-group comparisons (PG vs CAG) were calculated for the craniofacial starting forms at T1 and for the T2-T1 changes. Statistical between-group comparisons for the T2-T1 changes were performed with independent samples t-tests. The significance level was set at P <0.05. All statistical computations were performed with SPSS software (Statistical Package for the Social Sciences, SPSS, version 12, Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* bilateral Class II or end to end Class II molar relationship
* skeletal Class I or II malocclusion (ANB angle between 2° and 7°)
* normodivergence on the vertical plane (SN^GoGn angle less than 37°)
* crowding in the lower arch (≤6 mm)
* good quality of pre and post treatment radiographs
* good general health with healthy periodontium

Exclusion Criteria:

* patients who required functional appliance therapy
* those who had previous orthodontic treatment or extraction
* hypodontia
* craniofacial syndromes or cleft
* previous prosthodontic treatments of the upper molars

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
SN^GoGn | At the beginning and at the end of the teraphy
  The SN-GoGn angle is an angular measurement included in the study to quantify the inclination of the mandibular base relative to the cranial base. Its average value is 32°

SECONDARY OUTCOMES:
Overjet | At the beginning and at the end of the teraphy
  extension of the incisal or buccal cusp ridges of the upper teeth horizontally (labially or buccally) beyond the ridges of the teeth in the lower jaw when the jaws are closed normally.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome "Tor Vergata", Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Byloff FK, Darendeliler MA. Distal molar movement using the pendulum appliance. Part 1: Clinical and radiological evaluation. Angle Orthod. 1997;67(4):249-60. doi: 10.1043/0003-3219(1997)0672.3.CO;2. PMID 9267573
- [Background] Ghosh J, Nanda RS. Class II, Division 1 malocclusion treated with molar distalization therapy. Am J Orthod Dentofacial Orthop. 1996 Dec;110(6):672-7. doi: 10.1016/s0889-5406(96)80046-1. PMID 8972815
- [Background] Ravera S, Castroflorio T, Garino F, Daher S, Cugliari G, Deregibus A. Maxillary molar distalization with aligners in adult patients: a multicenter retrospective study. Prog Orthod. 2016;17:12. doi: 10.1186/s40510-016-0126-0. Epub 2016 Apr 18. PMID 27041551
- [Background] Angelieri F, de Almeida RR, Janson G, Castanha Henriques JF, Pinzan A. Comparison of the effects produced by headgear and pendulum appliances followed by fixed orthodontic treatment. Eur J Orthod. 2008 Dec;30(6):572-9. doi: 10.1093/ejo/cjn060. PMID 19054813
- [Background] de Almeida-Pedrin RR, Henriques JF, de Almeida RR, de Almeida MR, McNamara JA Jr. Effects of the pendulum appliance, cervical headgear, and 2 premolar extractions followed by fixed appliances in patients with Class II malocclusion. Am J Orthod Dentofacial Orthop. 2009 Dec;136(6):833-42. doi: 10.1016/j.ajodo.2007.12.032. PMID 19962606
- [Background] Hilgers JJ. The pendulum appliance for Class II non-compliance therapy. J Clin Orthod. 1992 Nov;26(11):706-14. No abstract available. PMID 1298751
- [Background] Bussick TJ, McNamara JA Jr. Dentoalveolar and skeletal changes associated with the pendulum appliance. Am J Orthod Dentofacial Orthop. 2000 Mar;117(3):333-43. doi: 10.1016/s0889-5406(00)70238-1. PMID 10715093
- [Background] Kravitz ND, Kusnoto B, BeGole E, Obrez A, Agran B. How well does Invisalign work? A prospective clinical study evaluating the efficacy of tooth movement with Invisalign. Am J Orthod Dentofacial Orthop. 2009 Jan;135(1):27-35. doi: 10.1016/j.ajodo.2007.05.018. PMID 19121497
- [Background] Rossini G, Parrini S, Castroflorio T, Deregibus A, Debernardi CL. Efficacy of clear aligners in controlling orthodontic tooth movement: a systematic review. Angle Orthod. 2015 Sep;85(5):881-9. doi: 10.2319/061614-436.1. Epub 2014 Nov 20. PMID 25412265
- [Background] Caruso S, Nota A, Ehsani S, Maddalone E, Ojima K, Tecco S. Impact of molar teeth distalization with clear aligners on occlusal vertical dimension: a retrospective study. BMC Oral Health. 2019 Aug 13;19(1):182. doi: 10.1186/s12903-019-0880-8. PMID 31409348
- [Derived] Lione R, Balboni A, Di Fazio V, Pavoni C, Cozza P. Effects of pendulum appliance versus clear aligners in the vertical dimension during Class II malocclusion treatment: a randomized prospective clinical trial. BMC Oral Health. 2022 Oct 10;22(1):441. doi: 10.1186/s12903-022-02483-w. PMID 36217134